CLINICAL TRIAL: NCT00873795
Title: Efficacy and Safety of Aripiprazole 2.5mg Combine Sertraline 50mg in Major Depression
Brief Title: Compare the Efficacy and Tolerability of the Combination of Aripiprazole and Selective Serotonin Reuptake Inhibitors (SSRIs) Used in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Fong-Lin Jang, Chi Mei Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 09603-001
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-04

CONDITIONS: Major Depressive Disorder
Keywords: efficacy; tolerability; combination of aripiprazole and SSRI(sertraline)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aripiprazole; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aripiprazole and sertraline (Experimental): The patients of this arm receive ten weeks of treatment with a combination of sertraline 50mg/day and aripiprazole 2.5mg/day.The effect of this arm is assessed for HAM-D17, CGI, SF-36 and BSRS-50.
  Interventions: Drug: aripiprazole , sertraline
- sertraline and placebo (Placebo Comparator): The patients of this arm receive ten weeks of treatment with a combination of sertraline 50mg/day and placebo.The effect of this arm is assessed for HAM-D17, CGI, SF-36 and BSRS-50.
  Interventions: Drug: aripiprazole , sertraline

INTERVENTIONS:
Drug: aripiprazole , sertraline — In this ten weeks,double-blind,placebo-control,randomized,fixed dose study, study,subjects were randomly assigned to treatment with aripiprazole 2.5mg/day plus sertraline 50mg/day or sertraline 50mg/day plus placebo.

SUMMARY:
FDA has accepted atypical antipsychotics of olanzapine and aripiprazole as the adjuvant medications for refractory major depression. But there is still no trial about atypical antipsychotics combined with antidepressant of SSRI used in fresh major depressive patients. This project aims to compare the efficacy and tolerability of sertraline with or without low-dosed aripiprazole added in fresh major depression.

DETAILED DESCRIPTION:
This double-blind, placebo-control, fixed dose, randomized study will be conducted at a tertiary clinical setting. Patients over 18 y/o fulfilled DSM-IV criteria for major depression, having a baseline HAM-D score ≧ 14 and a HAM-D item 3 score < 3 will be recruited into the groups. The study group of patients will receive ten weeks of treatment with a combination of fix-dosed sertraline and aripiprazole. The control group will received sertraline only. The score reduction in HAM-D17, CGI, SF-36 and Brief Symptom Rating Scale (BSRS-50) will be periodically estimated as an efficacy following the use of a SSRIs or and aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 65 years inclusive.
* Fulfilled DSM-Ⅳ criteria for major depressive disorder.
* Onset ≧2 weeks.
* Baseline score ≧14 on the HAM-D17.
* Written informed consent prior to entry into the study.

Exclusion Criteria:

* HAM-D17 item 3 score≧3.
* Life-time history of bipolar disorders, schizophrenia or schizoaffective disorder.
* Current history of panic disorder, obsessive-compulsive disorder, alcohol or substance abuse.
* Mood disorder due to general medical condition.
* Treatment with antidepressants at entry into the study before 2 weeks.
* Need for psychoactive medications other than the study drugs, except for one benzodiazepine or hypnotic given at a stable dose.
* Known intolerance or inefficacy to either drug.
* Previous lack of response to two or more antidepressants at adequate dosage.
* Subjects who have acute or unstable medical illness or organic failure.
* Pregnancy and breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
score change of Hamilton Rating Scale For Depression (HAM-D17 ) | day 1 / 1 week / 2 weeks/ 4 weeks/ 6 weeks/ 10weeks

SECONDARY OUTCOMES:
score change of Brief Psychiatric Rating Scale (BPRS-50) | day 1/ 1 week / 2 weeks/ 4 weeks/ 6 weeks/ 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Lin Jang, M.D., Study Director — Chimei Medical Center
Locations (1):
- Psychiatry Department, Chimei Medical Center, Tainan, Taiwan